CLINICAL TRIAL: NCT04277572
Title: Outcomes of Different Modalities for Surgery of Aortic Valve
Brief Title: Outcomes of Surgery of Aortic Valve
Acronym: Aortic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Thabet Ahmed, Assistant lecturer, Assiut University
Other Study IDs: 17200395
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aortic valve replacement: using different ways of aortic valve replacement either by prosthetic valves or by ozaki technique
  Interventions: Procedure: Aortic valve replacement

INTERVENTIONS:
Procedure: Aortic valve replacement — Aortic valve surgery
  Other Names: Ozaki procedure

SUMMARY:
Overall Goal: To study the outcomes of patients undergoing aortic valve surgeries, different approaches such as standard aortic valve replacement, aortic valve repair, novel techniques as Ozaki's procedure and their subsequent results and complications.

* Objective 1: Identify predictors of complications following different types of aortic valve surgery accordingly.
* Objective 2: Determine the value of each type in terms of advantages and disadvantages.
* Objective3: Assess outcomes such as postoperative life expectancy, hospital stay, prognosis and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe symptomatic aortic valve lesion.
2. Asymptomatic aortic insufficiency patients with left ventricular dysfunction or significant left ventricular dilatation (LV end diastolic diameter>70 mm or LV end systolic diameter>50 mm.
3. Patients with aortic regurgitation caused by:

   * a dilated aortic annulus
   * conjoined cusp prolapse in bicuspid aortic valves (BAV)
   * single cusp prolapse in tricuspid aortic valves
   * aortic valve cusp perforation from endocarditis

Exclusion Criteria:

* Patients with previous aortic root or valve surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered in cardiac surgery department database, and who meet the listed inclusion and exclusion criteria will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcomes of different techniques of aortic valve surgery in the indicated patients for each type of surgery such as : | Up to one week
  Number of days of postoperative hospital stay.

IPD SHARING:
Plan to Share IPD: No